CLINICAL TRIAL: NCT03372538
Title: is There Any Superior Benefit of Multidisciplinary Team in Management of Placenta Accreta
Brief Title: Multidisciplinary Team in Management of Placenta Accreta
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, sarah mohamed hassan, lecturer of obstetrics and gynecology, Kasr El Aini Hospital
Other Study IDs: 494608
Record Dates: First submitted 2017-12-09; First posted 2017-12-13 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Placenta Accreta
Keywords: placenta accreta
MeSH Terms: conditions — Placenta Accreta | interventions — Cesarean Section

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- multidisciplinary team group: 500 patients of placenta accreta managed by obstetricans and urologists
  Interventions: Procedure: cesarean section or cesarean hysterectomy
- obstetricians only group: 500 patients of placenta accreta managed by obstetricans only
  Interventions: Procedure: cesarean section or cesarean hysterectomy

INTERVENTIONS:
Procedure: cesarean section or cesarean hysterectomy — upper segment cesarean section and or cesarean hysteroctomy

SUMMARY:
comparative study between the incidence of urological injury in case of placenta accreta in cases where urological surgical staff are participating in the operation from the start and in cases where the operation is carried by the gynecological staff only

DETAILED DESCRIPTION:
cohort of 1000 patients of placenta accreta are followed regarding the incidence of urological injury in the cases with assistance from the urological staff members

ELIGIBILITY:
Inclusion Criteria:

* pregnant 38 weeks
* placenta accreta

Exclusion Criteria:

* medical disorders complicating pregnancy

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 1000 patients pregnant 38 weeks with placenta accreta
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-12 (Estimated); Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
urological injury | intraoperative
  badder or ureteric injury

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr El Ainiy Hospital, Cairo, Egypt